CLINICAL TRIAL: NCT02441465
Title: A Phase 1, Open-Label, Absolute Bioavailability Study of Vemurafenib in Patients With BRAF^V600 Mutation-Positive Malignancies
Brief Title: Bioavailability Study of Vemurafenib in Participants With BRAF^V600 Mutation-Positive Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GO28395; 2013-004144-34 (EudraCT Number)
Record Dates: First submitted 2015-04-30; First posted 2015-05-12 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Malignant Melanoma, Cancer
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vemurafenib (Experimental): Participants will receive oral vemurafenib BID from Day 1 to Day 28 and a single IV infusion of 14C-labeled vemurafenib on Day 21.
  Interventions: Drug: Vemurafenib; Drug: 14C-Labeled Vemurafenib

INTERVENTIONS:
Drug: Vemurafenib — Oral vemurafenib will be administered at a dose of 960 milligrams BID from Day 1 to Day 28.
  Other Names: Zelboraf®, RO5185426
Drug: 14C-Labeled Vemurafenib — IV infusion of 18.5 kilobecquerel (kBq) of 14C-labeled vemurafenib (3 milliliters [mL], which corresponds to a dose of 20 micrograms [mcg] of vemurafenib) on Day 21 (immediately after the morning oral dose of vemurafenib).

SUMMARY:
The purpose of this study is to characterize the pharmacokinetics (PK) of a single intravenous (IV) infusion of 14C-labeled vemurafenib administered shortly after an oral dose of vemurafenib and following multiple oral doses of vemurafenib twice daily (BID) at steady state as well as to estimate the absolute bioavailability of multiple oral doses of vemurafenib BID at steady state in participants with BRAF^V600 mutation-positive malignancies. The study has two periods: Period A and Period B. During Period A, participants will receive vemurafenib BID orally from Day 1 to Day 20 and during Period B, participants will receive single IV infusion of 14C-labeled vemurafenib along with vemurafenib BID oral dose.

ELIGIBILITY:
Inclusion Criteria:

* Participants with either unresectable or metastatic melanoma positive for the BRAF^V600 mutation or other malignant tumor type that harbors a V600-activating mutation of BRAF, and for whom vemurafenib is an accepted standard of care or where there is no other generally accepted standard of care
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Life expectancy greater than or equal to (>/=) 12 weeks
* Full recovery from the effects of any major surgery or significant traumatic injury within 14 days from the first dose of study drug
* Adequate hematologic and end organ function as defined by laboratory results obtained within 2 weeks prior to administration of study drug on Day 1
* Female participants of childbearing potential and male participants with partners of childbearing potential must agree to use two effective methods of contraception during the study and at least 6 months after completion of the study drug
* Negative serum pregnancy test results within 7 days prior to Day 1 in women of childbearing potential
* Absence of any psychological, familial, or sociological condition, or geographical constraints that could potentially hamper compliance with the study protocol and follow-up schedule

Exclusion Criteria:

* Prior anti-cancer therapy before the administration of study drug on Day 1
* Invasive malignancy other than BRAF mutant melanoma or other qualifying malignant tumor with BRAF^V600 mutation within the past 5 years
* History of clinically significant cardiac or pulmonary dysfunction
* Active central nervous system lesions
* Current, severe, uncontrolled systemic disease
* Inability or unwillingness to swallow tablets
* History of malabsorption, stomach or intestinal surgery/resection, or other condition that would potentially alter absorption and/or excretion of orally administered drugs
* History of clinically significant liver disease
* Active autoimmune disease
* Uncontrolled ascites requiring weekly large-volume paracentesis for 3 consecutive weeks prior to enrollment
* Pregnancy, lactation, or breastfeeding
* Need to take a concomitant medication, dietary supplement, or food that is prohibited during the study
* Known allergy or sensitivity to components of the vemurafenib formulation
* Active, uncontrolled or chronic infection requiring chronic suppressive antibiotics
* Use of any prescription medications/products, that are known to be strong cytochrome P450 (CYP)3A4 inhibitors or inducers within 2 weeks prior to Day 1
* Participation in any other investigational drug study in which receipt of an investigational study drug occurred within 30 days prior to Day 1 or within 5 times the elimination half-life of the respective drug (whichever is shorter)
* Participation in a trial involving administration of 14 C-radiolabeled compound(s) within 6 months prior to Day 1
* Poor peripheral venous access
* Any other acute or chronic condition that, in the opinion of the investigator, could limit the participant's ability to complete and/or participate in this clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-08-13 (Actual); Primary Completion 2016-08-18 (Actual); Study Completion 2017-01-09 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve (AUC) of 14C-Labeled Vemurafenib From Time 0 to Last Measurable Concentration Timepoint (AUC0-last) | Day 21: Predose (Hour 0); end of infusion (infusion duration: 15 minutes); 5, 15 and 30 minutes post-infusion; 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 168 hours post-infusion of 14C-labeled vemurafenib
AUC of 14C-Labeled Vemurafenib From Time 0 to Infinity (AUC0-inf) | Day 21: Predose (Hour 0); end of infusion (infusion duration: 15 minutes); 5, 15 and 30 minutes post-infusion; 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 168 hours post-infusion of 14C-labeled vemurafenib
AUC of Unlabeled Vemurafenib During the Dosing Interval (AUCtau) | Predose (0 hour) on Days 18, 19, 20; Day 21: pre-dose (0 hour), 15 minutes after oral dose (at the end of IV infusion), at 30 and 45 minutes, and 1.15, 2.25, 3.25, 4.25, 6.25, 8.25, and 12 hours following oral administration of unlabeled vemurafenib
Maximum Observed Plasma Concentration (Cmax) of 14C-Labeled Vemurafenib | Day 21: Predose (Hour 0); end of infusion (infusion duration: 15 minutes); 5, 15 and 30 minutes post-infusion; 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 168 hours post-infusion of 14C-labeled vemurafenib
Terminal Half-Life (t1/2) of 14C-Labeled Vemurafenib | Day 21: Predose (Hour 0); end of infusion (infusion duration: 15 minutes); 5, 15 and 30 minutes post-infusion; 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 168 hours post-infusion of 14C-labeled vemurafenib
Clearance (CL) of 14C-Labeled Vemurafenib | Day 21: Predose (Hour 0); end of infusion (infusion duration: 15 minutes); 5, 15 and 30 minutes post-infusion; 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 168 hours post-infusion of 14C-labeled vemurafenib
Volume of Distribution (V) of 14C-Labeled Vemurafenib | Day 21: Predose (Hour 0); end of infusion (infusion duration: 15 minutes); 5, 15 and 30 minutes post-infusion; 1, 2, 3, 4, 6, 8, 12 hours post-infusion of 14C-labeled vemurafenib
Absolute Bioavailability (%F) of Vemurafenib | Day 21 (detailed timeframe is provided in description field)
  %F is the ratio of dose normalized AUCtau following vemurafenib oral dose to dose normalized AUC0-inf following IV dose.
  Time Frame: Vemurafenib oral dose (Day 21: Predose [0 hour]; 15 minutes after oral dose [at the end of IV infusion], at 30 and 45 minutes, and 1.15, 2.25, 3.25, 4.25, 6.25, 8.25, and 12 hours following oral administration of unlabeled vemurafenib); Vemurafenib IV dose (Day 21: Predose [Hour 0]; end of infusion [infusion duration: 15 minutes]; 5, 15 and 30 minutes post-infusion; 1, 2, 3, 4, 6, 8, 12 hours post-infusion of 14C-labeled vemurafenib).
Renal Clearance (CLr) of 14C-Labeled Vemurafenib | Day 21 (urine samples): Predose (-8 to 0 hour), 0-4, 4-12, 12-24, 24-48, 48-72, 72-96 hours post-infusion (infusion duration: 15 minutes) of 14C-labeled vemurafenib
Total Amount of 14C-Labeled Vemurafenib (Parent Drug) Excreted Into Urine | Day 21 (urine samples): Predose (-8 to 0 hour), 0-4, 4-12, 12-24, 24-48, 48-72, 72-96 hours post-infusion (infusion duration: 15 minutes) of 14C-labeled vemurafenib

SECONDARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to 6 months after last dose (up to approximately 7 months)
Cmax of Unlabeled Vemurafenib | Predose (0 hour) on Days 18, 19, 20; Day 21: pre-dose (0 hour), 15 minutes after oral dose (at the end of IV infusion), at 30 and 45 minutes, and 1.15, 2.25, 3.25, 4.25, 6.25, 8.25, and 12 hours following oral administration of unlabeled vemurafenib
Time to Maximum Concentration (Tmax) of Unlabeled Vemurafenib | Predose (0 hour) on Days 18, 19, 20; Day 21: pre-dose (0 hour), 15 minutes after oral dose (at the end of IV infusion), at 30 and 45 minutes, and 1.15, 2.25, 3.25, 4.25, 6.25, 8.25, and 12 hours following oral administration of unlabeled vemurafenib
Percentage of 14C-Labeled Vemurafenib Dose Recovered as Total Radioactivity in Urine | Day 21 (urine samples): Predose (-8 to 0 hour), 0-4, 4-12, 12-24, 24-48, 48-72, 72-96 hours post-infusion (infusion duration: 15 minutes) of 14C-labeled vemurafenib
Percentage of 14C-Labeled Vemurafenib Dose Recovered as Total Radioactivity in Feces | Day 21 (feces samples): Predose (-48 to 0 hour), 0-24, 24-48, 48-72, 72-96, 96-120, 120-144, 144-196 hours post-infusion (infusion duration: 15 minutes) of 14C-labeled vemurafenib
14C-Labeled Vemurafenib Concentration Over Time Intervals in Urine | Day 21 (urine samples): Predose (-8 to 0 hour), 0-4, 4-12, 12-24, 24-48, 48-72, 72-96 hours post-infusion (infusion duration: 15 minutes) of 14C-labeled vemurafenib
14C-Labeled Vemurafenib Concentration Over Time Intervals in Feces | Day 21 (feces samples): Predose (-48 to 0 hour), 0-24, 24-48, 48-72, 72-96, 96-120, 120-144, 144-196 hours post-infusion (infusion duration: 15 minutes) of 14C-labeled vemurafenib

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Magyar Honvedseg Egeszsegugyi Kozpont, Budapest, Hungary